CLINICAL TRIAL: NCT00717899
Title: The Effect of Air Pollution on Lung Health Among School Children Living in Haifa Bay Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Haim Bibi, MD, Carmel Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HTA 4642/ CMC 0064-07; 3000004504 (Grant) (Other Grant/Funding Number: 3000004504)
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Bronchial Asthma; Signs and Symptoms, Respiratory; Allergy
Keywords: Asthma; Allergy; Respiratory; Pollution; Children; Air pollution
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory; Hypersensitivity | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): School children from Haifa bay region, Israel.
  Interventions: Device: Spirometry (Pony spirometer)

INTERVENTIONS:
Device: Spirometry (Pony spirometer) — Spirometry at rest
  Other Names: Pony spirometer, Cosmed, Italy

SUMMARY:
Haifa bay region is located close to a major industrial zone. The aim of the study is to evaluate the health status of school children living in Haifa bay region.The health status will be evaluated using health questionnaires and spirometry.

DETAILED DESCRIPTION:
Haifa bay is located close to a major industrial zone. The aim of the study is to evaluate the health status of children living in Haifa bay region.

The health status will be evaluated while using health questionnaires and spirometry.

Objective: To evaluate the respiratory health of Haifa bay region children with comparatives, with respect to local air pollution levels.

Material and Methods: Children from Haifa bay region from 10 different communities (1200 children) will be included in the study, after both parents and the children (above 12 years of age) will sign an informed consent form.

First step: A health questionnaire (based on Hebrew version of ISAAC questionnaire) will be filled in by the parents.

Second step: Spirometry checking of the children. In parallel, air pollution levels will be measured and provided by a network of ground monitoring stations maintained by the Haifa District Municipality Association for the Environment (HDMAE). The station provides half-hourly measurement of mean concentrations of gaseous (NOX, SO2, O3) and particular (PM 10) pollutants over the entire investigation window. Additional meteorological data are also collected.

Risk maps: Using a GIS platform, we are developing a multi-layer risk mapping procedure which accounts for ambient concentrations of selected pollutants and the heterogenic spatial distribution of several demographic and socio-economic indexes in the region.

The prevalence of pulmonary disease will be evaluated according to the risk maps The health status of the children will be documented from the children's primary clinic files as well.

ELIGIBILITY:
Inclusion Criteria:

* Living in Haifa bay region, Israel.
* Parents signed informed consent.

Exclusion Criteria:

* Children that their parents did not signed the informed consent
* Chronic disease except of asthma: Diabetes mellitus, Cystic Fibrosis, Cardiac diseases, Renal, Rheumatic and Chronic Gastrointestinal diseases, Mental retardation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The prevalence of respiratory symptoms in respect to air pollution | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Haim Bibi, MD, Principal Investigator — Carmel Medical Center, Haifa, Israel
Locations (1):
- Schools at the Haifa Bay region, Israel., Haifa Bay, Israel

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/15060197?ordinalpos=6&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum